CLINICAL TRIAL: NCT03509792
Title: Preventing Intrusive Memories After Trauma Via a Simple Cognitive Intervention in the Hospital Emergency Department: "EKUT" (Enkel Kognitiv Uppgift Efter Trauma)
Brief Title: Simple Cognitive Task After Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Emily Holmes, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017/2215-31
Record Dates: First submitted 2018-03-05; First posted 2018-04-26 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Post-traumatic Stress Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple cognitive task (Experimental): A memory cue followed by playing the computer game "Tetris" on own smartphone. Options to engage in self-administered booster sessions after day 1.
  Interventions: Behavioral: Simple cognitive task
- Attention placebo (Placebo Comparator): Smartphone activity for same amount of time.
  Interventions: Behavioral: Attention placebo

INTERVENTIONS:
Behavioral: Simple cognitive task — A memory cue followed by playing the computer game "Tetris" on own smartphone. Options to engage in self-administered booster sessions after day 1.
  Arms: Simple cognitive task
Behavioral: Attention placebo — Smartphone activity for same amount of time.
  Arms: Attention placebo

SUMMARY:
This research study is designed to investigate the effects of a simple cognitive task (a memory cue following by playing the computer game "Tetris") on intrusive memories ("flashbacks") and other symptoms after a traumatic event. Patients presenting to a hospital emergency department soon after a traumatic event will be randomly allocated to either the simple cognitive task intervention or control. Participants will be followed up at one week and one month, and where possible 3 and 6 months. It is predicted that participants given the simple cognitive task intervention will develop fewer intrusive memories and less severe clinical symptoms than those who are not. This will inform the potential future development of a simple technique to prevent distressing psychological symptoms after a traumatic event. Implementation aspects in a new hospital context will also be explored. Patients use their smartphone for part of the intervention in the study.

DETAILED DESCRIPTION:
This is an explorative pilot study, which will guide the design of a future Randomised Controlled Trial. The main aim of the present study is not a statistical significance test, the results will be descriptive, and will include pilot analyses to obtain an estimate of effect size between groups of the current primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Experienced or witnessed a traumatic event resulting in admission to the emergency department for example a road traffic accident (as a driver, passenger, motorcyclist, cyclist or pedestrian)
* Met the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM5) criterion A for Post-Traumatic Stress Disorder (PTSD) ("The person was exposed to: death, threatened death, actual or threatened serious injury, or actual or threatened sexual violence" by "Direct exposure" or "Witnessing the trauma") )
* Can be seen in the emergency department within 6 hours after the traumatic event
* Report memory of the accident
* Fluent in Swedish
* Alert and orientated
* Have sufficient physical mobility use the intervention platform (their smartphone) to play a computer game or engage in other smartphone activities at the point of taking informed consent (i.e. sufficient use of hands).
* Willing and able to provide informed consent and complete study procedures
* Willing and able to be contacted following discharge to complete follow-up assessments
* Have access to an internet enabled smartphone
* in addition to point above "can be seen in the emergency department within 6 hours after the traumatic event", from mid May 2019, to also include patients presenting later to the emergency department if still within 72 hours of the event

Exclusion Criteria:

* Loss of consciousness of > 5 minutes
* Current intoxication
* Report a history of severe mental illness
* Current substance abuse or neurological condition
* Currently suicidal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Number of intrusive memories of traumatic event | Week 1
  Number of intrusive memories of traumatic event recorded by participants in a diary daily (morning, afternoon, evening and night) for 7 days

SECONDARY OUTCOMES:
Number of intrusive memories of traumatic event | 1 month
  Number of intrusive memories of traumatic event recorded by participants in a diary daily (morning, afternoon, evening and night) for 7 days
Impact of Event Scale - Revised (IES-R) Intrusion Subscale: Degree of subjective distress of post-trauma symptoms in the intrusion (re-experiencing) symptoms cluster | One week and 1, 3, and 6month follow-up
  Full scale is a 22-item self-report measure that assesses subjective distress after a traumatic events. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The IES-R yields a total score (ranging from 0 to 88) and subscale scores are calculated for the Intrusion, Avoidance, and Hyperarousal subscales summed. Higher scores indicate worse outcome. Our secondary outcome measure is the Intrusion subscale.
Hospital Anxiety and Depression Scale (HADS): Anxiety and depressive symptoms | One week 1, 3, and 6 month follow-up
  The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. Higher scores indicate worse severity.
Perceived Stress Scale (PSS) | 1 month follow-up
  Measures the perception of stress and the degree to which situations in one's life are appraised as stressful. The 14 items aims to assess how unpredictable, uncontrollable, and overloaded respondents find their lives. The items are rated on a 5-point scale ranging from 0 ("never") to 4 ("very often") and summed to a total score of 56. Seven items concerns positive experiences and are hence reversed in scoring. Higher scores indicate worse severity.
Work and Social Adjustment Scale (WSAS): Daily function | [One week and 1, 3, and 6 month follow-up]
  The Work & Social Adjustment Scale is a simple 5-item measure of general social impairment which grew out of a study of change during psychotherapy. The maximum score of the WSAS is 40, lower scores are better.

OTHER OUTCOMES:
Feedback Questionnaire about Participation | One week and 1, 3, and 6 month follow-up
  22 bespoke items including questions about study participation e.g. how burdensome was it to participate in the study?" rated on 9-point scale from 1 (never) to 9 (always); and those about what has happened since the study with a yes/no response e.g. have you had any psychological or medical treatment since our last contact; and items with a free text response field e.g. do you have any comments about what it was like to take part in the study.
Implementation feedback | Day 1, week 1, and 1, 3 and 6 month follow ups, through to study completion
  Observation and qualitative interviews with participants, study team and staff regarding implementation of the procedures
Credibility/expectancy questionnaire: Treatment credibility | Day 1
  5 item questionnaire (11 item scale from 0 to 10) that rates to what degree the participants finds the intervention credible. High scores indicate greater credibility. A free text response field about activities engaged in during the assigned condition.
Self Rated Health (SRH) rating | baseline, one week and 1, 3, and 6 month follow-up
  A single item measuring perceived health status on a seven-point scale (from very good to very bad). High scores indicate good outcomes.
Self rated Sleep ratings | baseline, one week and 1, 3, and 6 month follow-up
  Two self rated items: Item 1 measures the extent of being troubled by poor sleep in the last month on a 5 point scale (from not at all to very much), and item 2 measures the number of nights in the week with sleep problems on 5 point scale (from 0-1 to 5-7 nights). Each 5-point scale is reverse scored (0 - 4) then summed. Possible total scores ranges from 0 - 8, with higher values indicative of better sleep.
Adverse events | One week 1, 3, and 6 month follow-up
  Adverse events and potential side effects associated with intervention
Characteristics and sensory modality of intrusive trauma memories | One week and 1 month follow-up
  7 self rated bespoke items measuring characteristics and sensory modality of intrusive memories: 1 self rated question regarding the presence and the extent of each of 7 sensory modalities in the intrusive memories (visual, auditory, tactile, somatic, olfactory, taste, and other sensations) measured on a scale from 1 (none) to 5 (extreme). 3 self rated items measuring the level of distress, vividness or disruption (functional impairment) associated with the intrusions (11 point scales from 0 to 10). High scores indicate higher level of distress/vividness/disruption.
M.I.N.I 7.0.0 (Mini International Neuropsychiatric Interview version 7.0.0) - Section H. Posttraumatic stress disorder (PTSD) | 1, 3, and 6 month follow-up
  Section H of MINI 7.0.0 (a short symptom interview) will be assessed at follow-ups to assess current symptoms of posttraumatic stress disorder. Section H consists of a minimum of 1 and maximum of 19 items, which continue depending on response to previous question). Higher scores indicate worse symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Emily Holmes, Prof, Principal Investigator — Karolinska Institutet; Erik Andersson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Akuten Huddinge Sjukhus, Stockholm, Solna, Sweden

REFERENCES:
- [Result] Kanstrup M, Singh L, Goransson KE, Widoff J, Taylor RS, Gamble B, Iyadurai L, Moulds ML, Holmes EA. Reducing intrusive memories after trauma via a brief cognitive task intervention in the hospital emergency department: an exploratory pilot randomised controlled trial. Transl Psychiatry. 2021 Jan 11;11(1):30. doi: 10.1038/s41398-020-01124-6. PMID 33431807
- [Result] Kanstrup M, Rudman A, Goransson K, Andersson E, Lauri KO, Rapoport E, Sunnergard L, Bragesjo M, Andersson E, Iyadurai L, Holmes EA. Reaching people soon after a traumatic event: an exploratory observational feasibility study of recruitment in the emergency department to deliver a brief behavioral intervention via smartphone to prevent intrusive memories of trauma. Pilot Feasibility Stud. 2021 Oct 7;7(1):184. doi: 10.1186/s40814-021-00916-x. PMID 34620249